# Healthy Immigrant Community: Mobilizing the Power of Social Networks

NCT05136339

October 15, 2021





Name and Clinic Number

Approval Date: October 15, 2021 Not to be used after: October 14, 2022

**Study Title:** Healthy Immigrant Community

**IRB#:** 21-009339

Principal Investigator: Wieland, Mark L., M.D. and Sia, Irene G., M.D., and Colleagues

During this research, information about your health will be collected. Under Federal law called the Privacy Rule, health information is private. However, there are exceptions to this rule, and you should know who may be able to see, use and share your health information for research and why they may need to do so. Information about you and your health cannot be used in this research study without your written permission. If you sign this form, it will provide that permission. You will be given a copy of this form.

## Your health information may be collected from:

- Past, present, and future medical records.
- Research procedures, including research office visits, tests, interviews, and questionnaires.

## Your health information will be used and/or given to others to:

- Do the research.
- Report the results.
- See if the research was conducted following the approved study plan, and applicable rules and regulations.

## Your health information may be used or shared with:

- Mayo Clinic research staff involved in this study.
- Other Mayo Clinic staff involved in your clinical care
- Researchers involved in this study at other institutions.
- The sponsor(s) of this study and the people or groups hired by the sponsor(s) to help perform this research.
- The Mayo Clinic Institutional Review Board that oversees the research.
- Federal and State agencies (such as the Food and Drug Administration, the Department of Health and Human Services, the National Institutes of Health, and other United States agencies) or government agencies in other countries that oversee or review research.
- A group that oversees the data (study information) and safety of this research.

## How your information may be shared with others:

While taking part in this study, you will be assigned a code that is unique to you but does not include information that directly identifies you. This code will be used if your study information is sent outside of Mayo Clinic. The groups or individuals who receive your coded information will use it only for the purposes described in this consent form.





Name and Clinic Number

Approval Date: October 15, 2021 Not to be used after: October 14, 2022

If the results of this study are made public (for example, through scientific meetings, reports, or media), information that identifies you will not be used.

In addition, individuals involved in study oversight and <u>not</u> employed by Mayo Clinic may be allowed to review your health information included in past, present, and future medical and/or research records. This review may be done on-site at Mayo Clinic or remotely (from an off-site location). These records contain information that directly identifies you. However, the individuals will not be allowed to record, print, or copy (using paper, digital, photographic, or other methods), or remove your identifying information from Mayo Clinic.

### Is your health information protected after it has been shared with others?

Mayo Clinic asks anyone who receives your health information from us to protect your privacy; however, once your information is shared outside Mayo Clinic, we cannot promise that it will remain private and it may no longer be protected by the Privacy Rule.

#### **Your Rights and Permissions**

Participation in this study is completely voluntary. You have the right not to participate at all. Even if you decide to be part of the study now, you may change your mind and stop at any time. You do not have to sign this form, but if you do not, you cannot take part in this research study.

Deciding not to participate or choosing to leave the study will not result in any penalty. Saying 'no' will not harm your relationship with your own doctors or with Mayo Clinic.

If you cancel your permission for Mayo Clinic to use or share your health information, your participation in this study will end and no more information about you will be collected; however, information already collected about you in the study may continue to be used.

You can cancel your permission for Mayo Clinic to use or share your health information at any time by sending a letter to the address below:

Mayo Clinic
Office for Human Research Protection
ATTN: Notice of Revocation of Authorization
201 Building 4-60
200 1st Street SW
Rochester, MN 55905

Alternatively, you may cancel your permission by emailing the Mayo Clinic Research Subject Advocate at: <a href="mayo.edu">researchsubjectadvocate@mayo.edu</a>.





Name and Clinic Number

Approval Date: October 15, 2021 Not to be used after: October 14, 2022

Please be sure to include in your letter or email:

- The name of the Principal Investigator,
- The study IRB number and /or study name, and
- Your contact information.

Your permission for Mayo Clinic to use and share your health information lasts forever unless you cancel it. There is no expiration or end date related to the Sponsor's use of your health information received from Mayo Clinic as part of this study.





Name and Clinic Number

**Approval Date:** October 15, 2021 Not to be used after: October 14, 2022

Your signature documents your permission to use your protected health information for this research.

| | / / | : | AM/PM |
|---|---|---|---|
| Printed Name | Date | Time | |
| Signature | | | |
| (Participant Parent/Guardian i | funder 18 or Legally Authorized | Representative) | |

(Participant, Parent/Guardian if under 18 or Legally Authorized Representative)